CLINICAL TRIAL: NCT05993065
Title: Study of Hematocrit to Hemoglobin Ratio and Red Blood Cell Distribution Width in Polycythemia Vera and Secondary Erythrocytosis
Brief Title: Hematocrit to Hemoglobin Ratio and Red Blood Cell Distribution Width in Polycythemia Vera and Secondary Erythrocytosis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Gaber Mahmoud, Dr, Sohag University
Other Study IDs: HCT to Hb and RDW in PV
Record Dates: First submitted 2023-08-06; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- polycythemia vera: All patients aged 18 years and older who were newly diagnosed to have polycythemia vera between September 2014 and November 2022 at Sohag university hospital, department of internal medicine, hematology unit and hematology outpatient clinic.
- secondary erythrocytosis: Patients with secondary erythrocytosis will be included as controls and will be recruited from Sohag university hospital especially internal medicine department and chest department. Patients of chronic respiratory failure, congenital heart diseases, polycystic kidney and other causes recruited in this study to be compared to PV group as regards Hematocrit to Hemoglobin Ratio and Red Blood Cell Distribution Width

SUMMARY:
Polycythemia vera (PV), a hematological neoplasm characterized by excessive erythropoiesis due to Janus kinase 2 (JAK2)- activating mutations. On the other hand, patients with secondary polycythemia (SP), a disorder mostly caused by an increased red cell mass due to chronic hypoxia (i.e, pulmonary disorders and smoking) and erythropoietin-producing tumors (such as leiomyoma, hemangiomas, renal cysts and various carcinomas), are phenotypically slightly different and are usually considered to have significantly better outcomes.

Red blood cell distribution width (RDW) reflects the heterogeneity of red blood cell sizes (anisocytosis) and is routinely reported as a part of complete blood count by automated instruments in hematology laboratories.

DETAILED DESCRIPTION:
We will collect data about clinical manifestations at the time of diagnosis, history of thrombosis and investigations as complete blood picture, including Hematocrit and haemoglobin level, serum uric acid, JAK2V617F mutation status by real time PCR (Polymerase Chain Reaction), bone marrow aspiration and biopsy with reticulin stain.

Patients with secondary erythrocytosis will be included as controls and will be recruited from Sohag university hospital especially internal medicine department and chest department.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and older who were newly diagnosed to have polycythemia vera between September 2014 and November 2022 at Sohag university hospital, department of internal medicine, hematology unit and hematology outpatient clinic.

Exclusion Criteria:

* Patients were excluded if: (1) their disease was not newly diagnosed, (2) their disease met WHO criteria for chronic, acute myeloid leukemia or other myeloid neoplasms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with polycythemia vera who were diagnosed according to the WHO 2016 criteria, at Sohag university hospital, department of internal medicine, hematology unit and hematology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Hematocrit to Hemoglobin Ratio in Polycythemia Vera and Secondary Erythrocytosis | Patients will be collected from December 2022 to September 2023
  We will collect data about clinical manifestations at the time of diagnosis, history of thrombosis and investigations as complete blood picture, including Hematocrit and haemoglobin level, serum uric acid, JAK2V617F mutation status by real time PCR (Polymerase Chain Reaction), bone marrow aspiration and biopsy with reticulin stain.
  Patients with secondary erythrocytosis will be included as controls and will be recruited from Sohag university hospital especially internal medicine department and chest department.
Red Blood Cell Distribution Width in Polycythemia Vera and Secondary Erythrocytosis | Patients will be collected from December 2022 to September 2023
  We will collect data about clinical manifestations at the time of diagnosis, history of thrombosis and investigations as complete blood picture, including Red Blood Cell Distribution Width, serum uric acid, JAK2V617F mutation status by real time PCR (Polymerase Chain Reaction), bone marrow aspiration and biopsy with reticulin stain.
  Patients with secondary erythrocytosis will be included as controls and will be recruited from Sohag university hospital especially internal medicine department and chest department.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Gaber, Principal Investigator — Sohag University
Locations (1):
- Faculty of Medicine, Sohag, Egypt

REFERENCES:
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Wouters HJCM, Mulder R, van Zeventer IA, Schuringa JJ, van der Klauw MM, van der Harst P, Diepstra A, Mulder AB, Huls G. Erythrocytosis in the general population: clinical characteristics and association with clonal hematopoiesis. Blood Adv. 2020 Dec 22;4(24):6353-6363. doi: 10.1182/bloodadvances.2020003323. PMID 33351130
- [Background] Nguyen E, Harnois M, Busque L, Sirhan S, Assouline S, Chamaki I, Olney H, Mollica L, Szuber N. Phenotypical differences and thrombosis rates in secondary erythrocytosis versus polycythemia vera. Blood Cancer J. 2021 Apr 15;11(4):75. doi: 10.1038/s41408-021-00463-x. No abstract available. PMID 33859172
- [Background] Holik H, Krecak I, Gveric-Krecak V, Vucinic Ljubicic I, Coha B. Higher red blood cell distribution width might differentiate primary from secondary polycythemia: A pilot study. Int J Lab Hematol. 2021 Apr;43(2):e68-e71. doi: 10.1111/ijlh.13373. Epub 2020 Oct 27. No abstract available. PMID 33108020
- [Background] Bhatt VR. Secondary polycythemia and the risk of venous thromboembolism. J Clin Med Res. 2014 Oct;6(5):395-7. doi: 10.14740/jocmr1916w. Epub 2014 Jul 28. No abstract available. PMID 25110547
- [Background] McMullin MF, Harrison CN, Ali S, Cargo C, Chen F, Ewing J, Garg M, Godfrey A, S SK, McLornan DP, Nangalia J, Sekhar M, Wadelin F, Mead AJ; BSH Committee. A guideline for the diagnosis and management of polycythaemia vera. A British Society for Haematology Guideline. Br J Haematol. 2019 Jan;184(2):176-191. doi: 10.1111/bjh.15648. Epub 2018 Nov 27. No abstract available. PMID 30478826